CLINICAL TRIAL: NCT04050410
Title: Autonomic Determinants of Postural Tachycardia Syndrome (Acute Pilot Study 1)
Brief Title: Autonomic Determinants of POTS - Pilot1
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Andre' Diedrich, Research Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: VANDERBILT_IRB_190703; R56HL142583 (NIH)
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Postural Tachycardia Syndrome
Keywords: postural tachycardia syndrome; hyperadrenergic; moxonidine; sympatholytic; orthostatic symptoms; POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — moxonidine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled crossover
Who Masked: Participant, Investigator
Masking Description: Subject and investigator will be blinded. The randomization will be generated by the pharmacy. A staff member of the Autonomic Dysfunction Center who is not involved in the study will keep secretly the randomization blinding table for emergencies. Blinding will be broken for intermediate data analysis and in case of emergencies if necessary. The blinding will be broken at the end of statistical analysis for interpretation of results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moxonidine (Experimental): Patients will receive a single oral dose of moxonidine 0.4 mg.
  Interventions: Drug: Moxonidine
- Placebo (Placebo Comparator): Patients will receive a single oral dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxonidine — active drug given as 1 dose
  Other Names: Physiotens
  Arms: Moxonidine
Drug: Placebo — placebo pill given as 1 dose
  Other Names: inactive pill
  Arms: Placebo

SUMMARY:
Postural tachycardia syndrome (POTS) is a relatively common condition affecting mostly otherwise healthy young women. It is the cause of significant disability and an impairment in quality of life. These patients have high heart rate and symptoms during standing. Many of these patients are disabled and have a poor quality of life. The sympathetic nerves are part of the nervous system that helps to maintain normal blood pressures and heart rates during activities of daily life. The purpose of this study is to determine the importance of sympathetic activation as a cause of orthostatic symptoms. The investigators will assess the effects of a blood pressure medication (Moxonidine) on the symptoms during standing. Moxonidine lowers sympathetic activity. The investigators believe patients with high resting sympathetic activity might benefit from Moxonidine. It might reduce high heart rate and improve symptoms during standing. This study should help clinicians and the growing population of patients with POTS gain a better understanding of this disorder and find more personalized treatment.

DETAILED DESCRIPTION:
Postural tachycardia syndrome (POTS) is a relatively common condition affecting mostly otherwise healthy young women. It is the cause of significant disability and an impairment in quality of life of a magnitude comparable to patients with chronic obstructive pulmonary disease or congestive heart failure. It is characterized by sympathetic activation with an exaggerated orthostatic tachycardia that responds to low doses of beta-blockers. The underlying pathophysiology of this disorder and the nature of this sympathetic activation is not clear and is likely heterogeneous. In many patients this sympathetic activation could be an appropriate compensatory response to hypovolemia, deconditioning or partial neuropathy.

The investigators have identified a subset of patients in whom sympathetic activation appears to be a primary phenomenon. These patients are characterized by high central sympathetic outflow, as determined by muscle sympathetic nerve activity (MSNA) above the upper 95% confidence interval for the group. This "hyperadrenergic" phenotype is associated with a paradoxical increase in blood pressure on standing and exaggerated pressor response to the vasoconstrictive phase of the Valsalva maneuver, and clinical observations suggest they improve clinically when treated with central sympatholytics.

The investigators propose to test the hypothesis that there is a subset of POTS patients with a central sympathetic activation as the primary pathophysiology. In an acute double blind, placebo-controlled, randomized study, the investigators propose that administration of the central sympatholytic moxonidine will improve orthostatic symptoms and abnormalities in orthostatic hemodynamics, as well as sympathetic outflow.

ELIGIBILITY:
Inclusion Criteria:

* female/male subjects, age 18-55 years,
* criteria for postural tachycardia syndrome (POTS):

  1. a heart rate increase of ≥30 beats/min within 10 minutes of upright posture;
  2. lack of orthostatic hypotension (blood pressure fall ≥ 20/10 mmHg within 10 minutes of standing); and
  3. chronic symptoms during upright posture over at least 6 months, in the absence of any other acute cause.
* in the follicular phase of the menstrual cycle (day 5-13 of a 28-day cycle)
* POTS with primary central sympathetic activation (psPOTS) as defined as having resting muscle sympathetic nerve activity (MSNA) greater than or equal to 25 bursts/min
* able and willing to provide informed consent.

Exclusion Criteria:

* pregnancy,
* smoker,
* BMI>30 kg/m2,
* deconditioned status (if available VO2max<80% of predicted)
* unable to withdraw from medications known to affect autonomic function, blood pressure or blood volume
* systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathies, and autoimmune neuropathies.
* Arteriosclerotic disease of carotid artery. History of neck surgery.
* conditions associated with inflammatory processes, such as coronary artery disease, hypertension, smoking, hypercholesterolemia (or on statin therapy), rheumatoid arthritis, diabetes
* treatment with oral corticosteroids, current infections (e.g., urinary tract infection), or use of non-steroidal anti-inflammatory drugs
* other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Orthostatic Symptom Burden [delta (delta VOSS)] | after 30 min supine to after 15 min upright (delta VOSS), 2-3 hours after placebo or moxonidine intake [delta (delta VOSS)].
  VOSS is a validated questionnaire that consists of 9 items: mental clouding, blurred vision, shortness of breath, rapid heartbeat, tremulousness, chest discomfort, headache, lightheadedness, and nausea. Each item is scored on a 0 to 10 scale (with 0 reflecting absence of symptoms), and the change of the total scores (range: 0-90) from supine to upright postures (delta VOSS) will be used as a measure of orthostatic symptom burden. The primary outcome measure will be the difference in orthostatic symptom burden [delta (delta VOSS)] following placebo vs. moxonidine administration.

SECONDARY OUTCOMES:
Change in Orthostatic Change in Heart Rate [delta (delta HR)] | after 30 min supine to after 15 min upright (delta HR), 2-3 hours after placebo or moxonidine intake [delta (delta HR)].
  Difference in heart rate change from supine to upright postures (delta HR) following placebo vs. moxonidine administration.

CONTACTS AND LOCATIONS:
Overall Officials: André Diedrich, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No